CLINICAL TRIAL: NCT06376136
Title: An Evaluation of BAT 8010 for Injection in Combination With BAT 1006 in Locally Advanced or Metastatic Entities Safety, Tolerability, Pharmacokinetic Profile, and Initial Clinical Efficacy of the Tumor in Patients Multicenter, Open Phase Ib/IIa Clinical Study
Brief Title: A Multicenter Open Clinical Study of Safety, Tolerability, Pharmacokinetic Profile, and Initial Clinical Efficacy of BAT 8010 for Injection Combined With BAT 1006 in the Treatment of Locally Advanced or Metastatic Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bio-Thera Solutions (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BAT-8010+1006-001-CR
Record Dates: First submitted 2024-04-17; First posted 2024-04-19 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A/ Standard 3+3 2.1mg/kg of BAT8010 (Experimental): Drug: BAT8010, Dosage: 2.1mg/kg, Frequency: once every 3 weeks, Duration: 1year
  Interventions: Drug: BAT8010 for Injection
- B/ Standard 3+3 2.4mg/kg of BAT8010 (Experimental): Drug: BAT8010, Dosage: 2.4mg/kg, Frequency: once every 3 weeks, Duration: 1year
  Interventions: Drug: BAT8010 for Injection
- C/ Standard 3+3 2.7 mg/kg of BAT8010 (Experimental): Drug: BAT8010, Dosage: 2.7 mg/kg, Frequency: once every 3 weeks, Duration: 1year
  Interventions: Drug: BAT8010 for Injection
- Standard 3+3 15 mg/kg of BAT1006 (Experimental): Drug: BAT1006, Dosage: 15 mg/kg, Frequency: once every 3 weeks, Duration: 1year
  Interventions: Drug: BAT1006 for Injection

INTERVENTIONS:
Drug: BAT8010 for Injection — Intravenous
  Arms: A/ Standard 3+3 2.1mg/kg of BAT8010; B/ Standard 3+3 2.4mg/kg of BAT8010; C/ Standard 3+3 2.7 mg/kg of BAT8010
Drug: BAT1006 for Injection — Intravenous
  Arms: Standard 3+3 15 mg/kg of BAT1006

SUMMARY:
This study is a multicenter, open, exploratory Phase Ib/IIa clinical trial in humans The combination of BAT8010 and BAT1006 was administered in patients with locally advanced or metastatic solid tumors(HER-2 expression, including IHC3+, IHC2+/FISH+, and IHC2+/FISH- patients)Tolerance and PK characteristics, to explore the maximum tolerated dose (MTD) and provide recommendations for subsequent clinical studies Recommended dose (RP2D) and rational administration regimen, and preliminary evaluation of antitumor efficacy. There are two main studies In the first stage, the "3+3" dose escalation rule is proposed to explore the safety and tolerance of the drug Sex; The second stage selects the appropriate dose and administration according to the preliminary safety and efficacy results of the previous stage The drug regimen and tumor species were expanded to further explore the combination of BAT8010 and BAT1006 for injection，The safety and clinical effectiveness of drug administration provided the basis for the follow-up clinical study.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥18 years old, male and female, voluntarily sign informed consent;
2. Estimated survival ≥3 months as assessed by the investigators;
3. the Eastern UnitedStates Cancer Consortium (ECOG) physicalstatu sscore requirements of 0 to 1 points;
4. Included in the crowd:

   1. Dose escalation stage: Patients with HER-2 expression confirmed by histopathology and cytopathology (including IHC3+, IHC2+/FISH+ and IHC2+/FISH-) who have failed standard therapy or have no standard treatment options or are not suitable for standard therapy at this stage, The climbing stage includes but is not limited to breast cancer, stomach cancer, non-small cell lung cancer, biliary tract cancer, colorectal cancer, urothelial carcinoma, etc.
   2. Dose expansion phase: divided into 3 cohorts i. Cohort A: Patients with breast cancer with HER-2 expression (including IHC3+, IHC2+/FISH+ and IHC2+/FISH-) confirmed by histopathology and cytopathology after failure of standard treatment or no standard treatment regimen or unsuitable for standard treatment at this stage; ii. Cohort B: Patients with histopathologically confirmed and inoperable locally advanced or metastatic urothelial carcinoma, including urinary bladder, pelvis, ureter, and urethral origin with HER-2 expression (including IHC3+, IHC2+/FISH+, and IHC2+/FISH-); iii. Cohort C: patients with gastric adenocarcinoma (including gastroesophageal junction adenocarcinoma) with disease progression after standard therapy, or histologically or cytologically proven metastatic or unresectable locally advanced or metastatic HER-2 expression (including IHC3+, IHC2+/FISH+, and IHC2+/FISH-) who are intolerant to standard therapy;
5. the dose escalation phase must have an evaluable tumor lesion, and the dose expansion phase must have at least one measurable tumor lesion (according to RECIST 1.1 criteria);
6. Pregnant women must have a negative pregnancy test during the screening period, before first dosing, and on the first day of each cycle. Consent must be given to the use of effective contraceptive methods to prevent pregnancy. No egg donation. And willing to take effective contraceptive methods to prevent pregnancy after signing the informed consent until 90 days after the last dosing of the study.

Exclusion Criteria:

1. During previous treatment with HER2-targeted drugs such as trastuzumab or pertuzumab, T-DM1, vedicitumab or Enhertu, as well as topoisomerase I inhibitors (such as irinotecan), grade 3 aes (including but not limited to infusion reactions or allergic reactions) that were determined to be treaty-related or of unknown drug relationship, or L after treatment VEF < 50%;
2. Participants who had previously received doxorubicin with cumulative dose > 360 mg/m2 or equivalent anthracyclines;
3. Before the first administration of the investigational drug, AE (CTCAE5.0) caused by previous antitumor therapy still had grade 1, except for the following cases: a. Hair loss; b Pigmentation; c. Patients with distal toxicity caused by chemotherapy and radiotherapy who can not be further recovered by judgment;
4. primary central nervous system tumor or symptomatic central nervous system metastasis, meningeal metastasis or a history of epilepsy. Patients with asymptomatic or asymptomatic central nervous system metastases under clinical control or who have symptoms but are judged to be stable by the investigators can be included, provided that the following conditions are met :a. The clinical symptoms were stable ≥4 weeks before the first dose. b. Brain MRI enhancement showed no evidence of progression of central nervous system disease within 4 weeks prior to initial administration; c. Antiepileptic drugs, hormones and other drugs have been stopped ≥2 weeks before the first administration;
5. Major surgical procedures were performed within 28 days prior to the first use of the study drug, or if postoperative complications persist after 21 days;
6. Subjects who have had a severe infection within 4 weeks prior to first dosing, or who have any signs and symptoms of active infection within 2 weeks prior to first dosing;
7. Subjects who have not been treated or are being treated for tuberculosis, including but not limited to tuberculosis (those who have been treated with standardized anti-tuberculosis therapy and have been confirmed cured by the investigator), a history of immunodeficiency, including human immunodeficiency virus (HIV) infection, or other immunodeficiency diseases, or a history of organ transplantation;
8. there are infected with the following diseases: active hepatitis B virus infection [hepatitis B surface antigen (HBsAg) positive, and hepatitis B virus deoxyribonucleic acid (HBV-DNA) test >200 IU/ml or 103 copies /ml (or > the normal high value of the study center detection)]; Hepatitis C virus infection [HCV antibody and viral ribonucleic acid (HCV-RNA) test positive]; Treponema pallidum antibody positive and RPR positive;
9. Patients with symptomatic congestive heart failure (NYHA grade II to IV) or severe arrhythmias requiring treatment (12-lead ECG QTc extension of 450 ms [male], 470 ms [female]), myocardial infarction, unstable angina in the last 6 months. Except atrial fibrillation or paroxysmal supraventricular tachycardia;
10. Patients with a history of non-infectious pneumonia requiring glucocorticoid therapy or with current interstitial lung disease;
11. the presence of any other serious underlying medical conditions (e.g. Gilbert's syndrome, uncontrolled diabetes, uncontrolled hypertension, active gastric ulcers, uncontrolled seizures, cerebrovascular events, gastrointestinal bleeding, severe signs and symptoms of coagulation and coagulation disorders), psychiatric/psychological/family factors that the investigator determines may influence screening, treatment, and follow-up. Affect compliance or put patients at high risk for treatment-related complications;
12. The previous anti-tumor therapy (such as chemotherapy, endocrine therapy, targeted therapy, immunotherapy or tumor embolization, etc.) is less than 28 days from the first study (or if the half-life of the drug is 5 times shorter than 28 days, the sponsor and the researcher shall decide whether to include it according to the specific analysis of the specific circumstances). Note that castration for prostate cancer and bisphosphonate or dinomumab for osteoporosis are permitted. Patients whose previous palliative radiotherapy was less than 7 days removed from the first study, or whose previous wide-field radiotherapy was less than 28 days removed from the first study, or who had not recovered from the side effects of radiotherapy as determined by the investigators;
13. Therapeutic radiopharma use must be discontinued 8 weeks before the first study administration;
14. Known allergy or intolerance to the investigational drug or its excipients;
15. Pregnant or lactating women;
16. Subjects considered unsuitable for participation in this study by the researcher.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2024-05-08 (Actual); Primary Completion 2026-11-09 (Estimated); Study Completion 2026-12-09 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | The first administration cycle(21 days)
  DLT events and their incidence.
vital signs | Through study completion, 1 year
  Number of participants with abnormal vital signs
Physical examination | Through study completion, 1 year
  Number of participants with abnormal physical examination
Adverse events | From the first receipt of the investigational drug until 28 (+7) days after the last receipt of the investigational drug or the initiation of a new antitumor therapy, whichever occurs earlier，assessed up to 1 year
  Number of cases with all adverse medical events that occur after the subject receives the investigational drug
Clinical laboratory tests | Through study completion, 1 year
  Number of participants with abnormal Clinical laboratory tests
Number of participants with abnormal clinical auxiliary tests | Through study completion, 1 year
  Clinical auxiliary tests
Duration of Response(DOR) | Through study completion, 1 year
  DoR is defined as the time between the first assessment of objective remission of a tumor and death from any cause before the first assessment of Disease progression (PD) , reflecting the duration of ORR
Disease Control Rate (DCR) | Through study completion, 1 year
  The proportion of patients with tumor reduction or stability maintained for a certain period, including cases of complete response (CR), partial response (PR), and stable disease (SD)

SECONDARY OUTCOMES:
Pharmacokinetic | At the end of Cycle 1 Day 1 to Cycle 1 Day 4, Cycle 1 Day 8，Cycle 1 Day 15, Cycle 2 Day 1，Cycle 3 Day 1 to Cycle 3 Day 3 , Cycle 3 Day 8 , Cycle 3 Day 15，Cycle 4 Day 1 ,Cycle 5 Day 1 ，Cycle 6 Day 1，EOT until 17 cycles (one cycle equals 2 weeks)
  Level of Cmax
Pharmacokinetic | At the end of Cycle 1 Day 1 to Cycle 1 Day 4, Cycle 1 Day 8，Cycle 1 Day 15, Cycle 2 Day 1，Cycle 3 Day 1 to Cycle 3 Day 3 , Cycle 3 Day 8 , Cycle 3 Day 15，Cycle 4 Day 1 ,Cycle 5 Day 1 ，Cycle 6 Day 1，EOT until 17 cycles (one cycle equals 2 weeks)
  Level of Tmax
Pharmacokinetic | At the end of Cycle 1 Day 1 to Cycle 1 Day 4, Cycle 1 Day 8，Cycle 1 Day 15, Cycle 2 Day 1，Cycle 3 Day 1 to Cycle 3 Day 3 , Cycle 3 Day 8 , Cycle 3 Day 15，Cycle 4 Day 1 ,Cycle 5 Day 1 ，Cycle 6 Day 1，EOT until 17 cycles (one cycle equals 2 weeks)
  Level of CL
Pharmacokinetic | At the end of Cycle 1 Day 1 to Cycle 1 Day 4, Cycle 1 Day 8，Cycle 1 Day 15, Cycle 2 Day 1，Cycle 3 Day 1 to Cycle 3 Day 3 , Cycle 3 Day 8 , Cycle 3 Day 15，Cycle 4 Day 1 ,Cycle 5 Day 1 ，Cycle 6 Day 1，EOT until 17 cycles (one cycle equals 2 weeks)
  Level of T1/2
Antibody | At the end of Cycle 1 Day 1, Cycle 2 Day 1，Cycle 3 Day 1 ,Cycle 5 Day 1，Cycle 6 Day 1，EOT until 17 cycles (one cycle equals 2 weeks)
  Level of ADA
Antibody | At the end of Cycle 1 Day 1, Cycle 2 Day 1，Cycle 3 Day 1 ,Cycle 5 Day 1，Cycle 6 Day 1，EOT until 17 cycles (one cycle equals 2 week
  Level of Nab

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Xu, Principal Investigator — Medical Ethics Committee of Sun Yat-sen University Cancer Center
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China